CLINICAL TRIAL: NCT06325215
Title: The Impact of Hydrocolloid on Preventing Pressure Injuries in the Nose and Columella of Preterm Infants: " A Randomized Controlled Trial"
Brief Title: The Effect of Hydrocolloid to Prevent Nasal Injuries in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Caglar, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SCaglar
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pressure Injury
Keywords: nasal injuries; hidrocolloid tape; collumela; non-invasive mechanic ventilation; preterm infants
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimantal
Who Masked: Care Provider, Investigator
Masking Description: After providing information about the study to the parents of preterm newborns who met the inclusion criteria, informed consent forms were obtained without disclosing which group their babies would be assigned to. The research outcome measurements were recorded by two nurses working at NICU. Prior to the study, necessary training and information about the form and process were provided to the nurses. The data analysis was conducted by an independent statistician.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocolloid tape group (Experimental): In this group, after the columella and nasal area of preterm infants were cleaned and dried with sterile water, hydrocolloid dressings were applied to the areas in contact with the nasal cannula. NasalNem nasal ointment was applied twice a day to the nasal passages in contact with the cannula. If the hydrocolloid dressings melted or peeled off, they were removed, the area was cleaned, and then reapplied. In the data collection process, assessments of the included preterm infants were conducted by two nurses. The upper lip, nasal passages, nasal septum, and columella region of the preterm infants were evaluated.
  Interventions: Other: Hidrocolloid Bant
- Control group (No Intervention): In this group, premature infants underwent the routine procedure of the NICU. As per the clinic's routine procedure, after cleaning and drying the columella and nasal area with sterile water, NasalNem nasal ointment was applied twice a day to the nasal passages in contact with the cannula. In the data collection process, assessments of the included preterm infants were conducted by two nurses. The upper lip, nasal passages, nasal septum, and columella region of the preterm infants were evaluated.

INTERVENTIONS:
Other: Hidrocolloid Bant — In this group, after the columella and nasal area of preterm infants were cleaned and dried with sterile water, hydrocolloid dressings were applied to the areas in contact with the nasal cannula. NasalNem nasal ointment was applied twice a day to the nasal passages in contact with the cannula. If the hydrocolloid dressings melted or peeled off, they were removed, the area was cleaned, and then reapplied.
  Arms: Hydrocolloid tape group

SUMMARY:
The aim of this study is to evaluate the effect of using hydrocolloid tapes in preventing pressure injuries on the nose and columella regions caused by non-invasive mechanical ventilation (NIMV) in preterm infants.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of using hydrocolloid tapes in preventing pressure injuries on the nose and columella regions caused by non-invasive mechanical ventilation (NIMV) in preterm infants.

This study is a, prospective randomized controlled trial.The research population comprised 56 premature neonates born at 37 weeks of gestation or less, who received NIMV support in the neonatal intensive care unit (NICU) between May 2022 and November 2022. Participants were randomly assigned to one of two groups; the first group (n=28) received hydrocolloid band application, while the second group (n=28) served as the control group. "Data Collection Form", "Neonatal Skin Risk Assessment Scale (NSRAS)", "Neonatal Skin Condition Score (NSCS)" and "Pressure Injury Staging Scale (PISS)" were used for data collection.

Intervention Tools:

For the NIMV of premature infants, Alpha brand nasal cannulas were used. The nasal cannula has soft binasal tips and is suitable for both low and high flow oxygen usage. A new sterile cannula was used for each infant.

Abfen-Farma brand Nasalnem Nasal Ointment was used for premature infants. Nasalnem Nasal Ointment aids in healing wounds inside the nose, resolving problems such as mucosa regeneration and mucosal wounds, supporting the mucosa, and alleviating issues like crusting and dryness.

In the hydrocolloid barrier group, Hartmann brand hydrocolloid tape was used.Hydrocolloid tape is a type of dressing used in wound care, consisting of a flexible, water-resistant adhesive containing a gel-forming substance such as pectin, gelatin or cellulose. Hydrocolloid tapes create a moist environment by being applied directly onto the wound, which accelerates healing and helps prevent infection. The adhesive layer of the dressing forms a barrier that protects the wound from external contaminants while providing support and reducing friction. Hydrocolloid tapes are available in various shapes and sizes and have the ability to remain in place for several days without needing to be changed. This feature can be beneficial in terms of patients, caregivers and cost-effectiveness .

Hydrocolloid band group (n=28): In this group, after the columella and nose areas of preterm infants were cleaned and dried with sterile water, hydrocolloid bands were placed on the areas where the nasal cannula made contact. NasalNem nasal ointment was applied twice a day to the nasal passages in contact with the cannula. If the hydrocolloid bands melted or detached, they were removed, the area was cleaned, and then reapplied. The nose and columella regions of preterm infants were evaluated every 12 hours for a total of 4 days/96 hours using the NSRAS scale for skin risk status, the NSCS scale for dryness, redness and peeling status, and the PISS scale for the occurrence of pressure injuries.

Control group (n=28): Preterm infants in this group were subjected to the routine procedure of the NICU. According to the clinic's routine procedure, after cleaning and drying the columella and nose areas with sterile water, NasalNem nasal ointment was applied twice a day to the nasal passages in contact with the cannula. The nose and columella regions of preterm infants were evaluated every 12 hours for a total of 4 days/96 hours using the NSRAS scale for skin risk status, the NSCS scale for dryness, redness and peeling status and the PISS scale for the occurrence of pressure injuries.

ELIGIBILITY:
Inclusion Criteria:

* Were born at less than 37 weeks of gestation,
* Were admitted to the neonatal intensive care unit,
* Received non-invasive mechanical ventilation support for at least 4 days,
* Were approved for inclusion in the study by their families.

Exclusion Criteria:

* Have been intubated,
* Have congenital anomalies,
* Have a history of nasal trauma,
* Have skin diseases,
* Have sensitivity or allergies to hydrocolloid tape.

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Neonatal Skin Condition Score | every 12-hour shift over 4 days for assessment
  he measuring tool consists of three items, each with an assessment criterion. These are dryness, erythema, and skin integrity impairment/peeling, respectively. The first item; Dryness (1=Normal, no signs of dryness, 2= Dry skin, visible flaking, 3= Very dry skin, cracking/fissures), the second item; Redness (1= No signs of redness, 2= Visible redness in less than 50% of the body surface, 3= Visible redness in more than 50% of the body surface), the third item; Skin Integrity Impairment / Peeling (1= No signs, 2= Limited impairment/peeling in a small area, 3= Extensive impairment/peeling). Developed in a triple Likert scale format, each item of the scale receives scores from 1 (one) to 3 (three). The lowest score that can be obtained from the scale is 3, and the highest score is 9; with a high total score indicating poor skin condition in the newborn.
Pressure İnjury Staging Scale | every 12-hour shift over 4 days for assessment
  The scale consists of six stages:
  I. Stage: Non-blanchable erythema that does not fade with pressure on intact skin, II. Stage: Partial thickness loss of dermis and blistering, III. Stage: Loss involving full thickness of skin and subcutaneous tissue, IV. Stage: Full thickness tissue loss (bone/muscle visible), Unstageable / Unclassifiable Stage: Loss of all layers of skin or tissues (depth unknown), Suspected Deep Tissue Injury: Depth Unknown.

SECONDARY OUTCOMES:
Neonatal Skin Risk Assessment Scale | every 12-hour shift over 4 days for assessment
  This scale consists of six parameters specific to the newborn population (general physical condition, mental state, mobility, activity, nutrition, and moisture), and it is adjusted according to gestational age. Each parameter is scored from 1 to 4. The total score ranges from 6 to 24. A high score indicates an increased risk of skin integrity impairment in the newborn, whereas a low score indicates a low risk of skin integrity impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Abide-i Hurriyet Cad. Istanbul University-Cerrahpaşa, Florence Nightingale Faculty of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No